CLINICAL TRIAL: NCT03873753
Title: Relationship Between Oral Hygiene in Newborns and Candida Spp.: A Randomized Clinical Trial
Brief Title: Relationship Between Oral Hygiene in Newborns and Candida Spp.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Faculty Sao Leopoldo Mandic Campinas (Other)
Responsible Party: Principal Investigator, Jose Carlos P Imparato, PhD, Senior Lecturer, Clinical Professor, Faculty Sao Leopoldo Mandic Campinas
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SLM 6
Record Dates: First submitted 2019-02-21; First posted 2019-03-13 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Candidiasis, Oral
Keywords: Pediatric dentistry; Mouth, Edentulous
MeSH Terms: conditions — Candidiasis, Oral; Mouth, Edentulous

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral cleaning (Experimental): The oral cavity will be clean with gauze and mineral water three times a day.
  Interventions: Other: Cleaning
- No oral cleaning (Active Comparator): The oral cavity will not be cleaned.
  Interventions: Other: No oral cleaning

INTERVENTIONS:
Other: Cleaning — Gauze and mineral water
  Arms: Oral cleaning
Other: No oral cleaning — Absence of cleaning
  Arms: No oral cleaning

SUMMARY:
Little is known regarding the effectiveness of neonatal oral hygiene and its relationship to colonization by Candida spp. in edentulous oral cavities. Thus, the objective of this study is to evaluate whether the oral hygiene of edentulous infants favors colonization by Candida spp. Newborns with up to 48 hours of life will randomly allocated to two groups. The mothers will instructed to clean the oral cavity with gauze and mineral water three times a day, in the test group, and not to clean, in the control group.

ELIGIBILITY:
Inclusion Criteria:

* A signed statement of informed consent
* Newborns up to 48 hours of life
* Exclusive breastfeeding
* Edentulous oral cavity

Exclusion Criteria:

* Any feeding other than breastfeeding
* Use of pacifier
* Digit sucking
* Systemic alterations

Max Age: 2 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 276 (Estimated)
Dates: Start 2017-05-02 (Actual); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from number of Candida spp CFU/mm3 | At baseline as well as once a month until the eruption of the first tooth (up to 14 months)
  Non-stimulated saliva will be collected with the aid of a sterile swab (Absorve®) from all infants. The samples were incubated at 37°C and analyzed after 48 hours to quantify the colony forming units (CFU/mm3)

SECONDARY OUTCOMES:
Mean of patient's birth weight in the test group as assessed by questionnaire | At baseline as well as once a month until the eruption of the first tooth (up to 14 months)
Number of males in the test group as assessed by questionnaire | At baseline as well as once a month until the eruption of the first tooth (up to 14 months)
Number of cesarean delivery in the test group as assessed by questionnaire | At baseline as well as once a month until the eruption of the first tooth (up to 14 months)
Mean of patient's gestational week in the test group as assessed by questionnaire | At baseline as well as once a month until the eruption of the first tooth (up to 14 months)
Mean of patient's birth length in the test group as assessed by questionnaire | At baseline as well as once a month until the eruption of the first tooth (up to 14 months)

CONTACTS AND LOCATIONS:
Overall Officials: Jose Carlos P Imparato, PhD, Principal Investigator — Faculdade Sao Leopoldo Mandic, Campinas, SP, Brazil
Locations (1):
- Faculty Sao Leopoldo Mandic, Campinas, São Paulo, Brazil